CLINICAL TRIAL: NCT05421988
Title: Effectiveness of Group and Individual Training in Emotional Freedom Techniques for Patients in Remission From Melanoma
Brief Title: Effectiveness of Group and Individual Training in EFT for Patients in Remission From Melanoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: NIIH20220324
Record Dates: First submitted 2022-04-03; First posted 2022-06-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants in the two treatment arms, and data analysts, will be blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual EFT Therapy (Experimental): Personal EFT instruction and practice group
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)
- Group EFT Therapy (Experimental): Group EFT instruction and practice group
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)
- Wait List (No Intervention): Wait list control group

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques (EFT) — EFT is an efficacious method demonstrated in over 100 clinical trials. It combines cognitive and exposure techniques with acupressure, in the form of fingertip percussion on acupuncture meridian points.
  Arms: Group EFT Therapy; Individual EFT Therapy

SUMMARY:
Serious medical diagnosis frequently induce fear focused on specific anticipations or generalized anxiety, along with uncertainty, insecurity, and disorientation. Other emotions such as anger, depression, hopelessness, shame, or grief may also become involved following a serious diagnosis. The adverse impact of stress on health and immune function is well-established, as well as its link to depression and anxiety. Emotional Freedom Techniques (EFT) has demonstrated efficacy in treating anxiety, depression, and PTSD. This study tests its effectiveness in reducing negative emotional symptoms in general, and fear of recurrence in particular, among individuals previously diagnosed with melanoma and currently in remission.

DETAILED DESCRIPTION:
Serious medical diagnosis frequently induce fear focused on specific anticipations or generalized anxiety, along with uncertainty, insecurity, and disorientation. Other emotions such as anger, depression, hopelessness, shame, or grief may also become involved following a serious diagnosis. The adverse impact of stress on health and immune function is well-established, as well as its link to depression and anxiety. Emotional Freedom Techniques (EFT) has demonstrated efficacy in treating anxiety, depression, and PTSD. This study tests its effectiveness in reducing negative emotional symptoms in general, and fear of recurrence in particular, among individuals previously diagnosed with melanoma and currently in remission.

Specifically, the study aims:

1. To assess the effect of instruction and practice of EFT on illness perception, fear of cancer recurrence, and wellbeing.
2. To assess whether the social support provided by EFT instruction in a group setting makes this efficient mode of implementation non-inferior or even beneficial in comparison to personal instruction.
3. To describe the emotions related to life events reported by patients in connection with the appearance and location of melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma diagnosis over six months prior to the study; confirmed by clinical, dermoscopic examination and pathology results

Exclusion Criteria:

* In active treatment for melanoma
* schizophrenia
* epilepsy
* other malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Illness perception | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change in score on Revised Illness Perception Questionnaire (IPQ-R)
Perception of recurrence | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change of perceived recurrence risk on a Likert scale

SECONDARY OUTCOMES:
Other physical symptoms | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change in patient's self-report of somatization, pain, and other symptoms on a Likert scale
Depression | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change in depressive symptoms on the Positive and Negative Affect Schedule (PANAS)
Anxiety | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change in anxiety symptoms on the Positive and Negative Affect Schedule (PANAS)
Patient's self-report of quality of life | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change in quality of life scores on the Quality of Life Scale (QOLS)
Wellbeing | Pre intervention, post 4 week intervention, and 3 month follow-up
  Change in score on The Well-being Numerical Rating Scales (WB-NRSs).

CONTACTS AND LOCATIONS:
Overall Officials: Yael Benyamini, PhD, Study Director — Tel Aviv University
Locations (1):
- The School Of Social Work Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
An anonymized data file will be made available to any other qualified investigator who requests it.
Time Frame: Data will be made available upon publication and for 5 years thereafter.
Access Criteria: Email request from qualified investigator.

REFERENCES:
- [Derived] Lazarov A, Church D, Shidlo N, Benyamini Y. The Effectiveness of Group and Individual Training in Emotional Freedom Techniques for Patients in Remission from Melanoma: A Randomized Controlled Trial. Healthcare (Basel). 2025 Jun 13;13(12):1420. doi: 10.3390/healthcare13121420. PMID 40565447